CLINICAL TRIAL: NCT06964399
Title: Psychological Well-Being and Mindfulness in the Elderly: The Effect of Reminiscence Therapy
Brief Title: The Effect of Reminiscence Therapy in Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: Reminiscence Therapy
Record Dates: First submitted 2025-04-24; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Age-related Cognitive Decline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Reminiscence Therapy can be applied as 1 or 2 sessions per week and the longest is 1.5 hours, so it will be applied for 5 weeks, 3 days a week (Monday, Wednesday, Friday) with 2 sessions per day. Each session is planned to last an average of 1.5 hours according to the answers from the elderly. The elderly individuals in the experimental group will be divided into 3 groups. Each group will consist of 15 people. The sessions will include, respectively, getting to know each other, childhood, places lived, holidays-festivals, foods-cooking, unforgettable historical periods, favorite music, movies specific to the period, family life-values in life-achievements, evaluation and closing topics.
  Interventions: Other: Reminiscence therapy
- Control Group (No Intervention): There will be no intervention in the control group during the research process.

INTERVENTIONS:
Other: Reminiscence therapy — Reminiscence Therapy can be applied as 1 or 2 sessions per week and the longest is 1.5 hours, so it will be applied for 5 weeks, 3 days a week (Monday, Wednesday, Friday) with 2 sessions per day. Each session is planned to last an average of 1.5 hours according to the answers from the elderly. The elderly individuals in the experimental group will be divided into 3 groups. Each group will consist of 15 people. The sessions will include, respectively, getting to know each other, childhood, places lived, holidays-festivals, foods-cooking, unforgettable historical periods, favorite music, movies specific to the period, family life-values in life-achievements, evaluation and closing topics.
  Arms: Experimental Group

SUMMARY:
In this study titled "Psychological Well-Being and Awareness in the Elderly: The Effect of Reminiscence Therapy", patients will be randomly divided into two groups as experimental and control groups. No intervention will be made to the patients in the control group. Reminiscence therapy will be applied to the patients in the experimental group. Participants will be asked to fill out the scale forms after accepting to participate in the study and obtaining their consent. In addition, after the reminiscence therapy is completed, the experimental and control groups will be asked to fill out the post-test forms.

The following questions will be answered in the study;

* Does reminiscence therapy affect the psychological well-being levels of the elderly?
* Does reminiscence therapy affect the awareness levels of the elderly?

DETAILED DESCRIPTION:
With the aging society in the world and in our country, there is a great need for the development of nursing interventions that will improve and sustain the health and quality of life of the elderly, who are increasingly included in the service area of nurses. It is very important for nurses to perform non-pharmacological practices, which are among their independent functions, not only for the patient but also for their own professional satisfaction. In these services, complementary therapies related to strengthening the personal resources of elderly individuals and ensuring their correct use are important. Therefore, this study aimed to determine the effect of reminiscence therapy applied to elderly individuals on their psychological well-being and awareness levels. In this study titled "Psychological Well-being and Awareness in the Elderly: The Effect of Reminiscence Therapy", patients will be randomly divided into two groups as experimental and control groups. No intervention will be made to the patients in the control group. Reminiscence therapy will be applied to the patients in the experimental group. Participants will be asked to fill out the scale forms after accepting to participate in the study and obtaining their consent. In addition, after the end of the reminiscence therapy, the experimental and control groups will be asked to fill out the final test forms.

The following questions will be answered in the research;

* Does reminiscence therapy affect the psychological well-being levels of the elderly?
* Does reminiscence therapy affect the awareness levels of the elderly?

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years old
* not having any serious psychiatric disorders
* not having any diseases such as dementia etc.

Exclusion Criteria:

* Having a serious psychiatric disorder
* Not being able to attend sessions during the research process

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Psychological well-being Scale | 1 months
  scale score average, It is a single-factor scale consisting of 8 items on a 7-point Likert type. Scores range from 8 to 56. A high score obtained from the scale indicates that the person has many psychological resources and strengths.

CONTACTS AND LOCATIONS:
Overall Officials: Güzel Nur YILDIZ, Dr, Principal Investigator — Muş Alparslan University
Locations (1):
- Ağın Community Health Center, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No